CLINICAL TRIAL: NCT04561128
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Administered SHR-1819 in Healthy Subjects
Brief Title: A Trial of SHR-1819 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1819-I-101-AUS
Record Dates: First submitted 2020-08-29; First posted 2020-09-23 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1819 (Experimental): Experimental: SHR-1819
  Interventions: Drug: SHR-1819
- Placebo (Placebo Comparator): Placebo comparator: placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1819 — SHR-1819 will be subcutaneously administered with different dose levels
  Arms: SHR-1819
Drug: Placebo — Placebo will be subcutaneously administered with different dose levels
  Arms: Placebo

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, single dose escalation phase 1 study.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo-controlled, single dose escalation phase 1 study. The objective of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of subcutaneous administered SHR-1819 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial, and provides written informed consent.
* Be able to comply with all the requirements and able to complete the study.
* Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
* No clinically significant abnormalities in medical history, general physical examination, vital signs, and laboratory tests.
* Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods and have no plan to have a child from signing the consent form to 16 weeks after IP administration.

Exclusion Criteria:

* Positive hepatitis B virus (HBsAg), hepatitis C virus (HCV-Ab), human immunodeficiency virus (HIV-Ab), or QuantiFERON-TB Gold tests at screening;
* Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening (according to the date of signed consent form), or in the follow-up period of a clinical study
* Severe injuries or surgeries within 6 months before screening or plan to do surgeries during the trial
* Any other circumstances that, in the investigator's judgment, may increase the risk associated with the subject's participation in and completion of the study or could preclude the evaluation of the subject's response

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 13 weeks)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 13 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1819 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 13 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1819 administration
Pharmacokinetics-Tmax | Up to 13 weeks
  Time to Cmax of SHR-1819
Pharmacokinetics-Cmax | Up to 13 weeks
  Maximum observed concentration of SHR-1819
Pharmacokinetics-CL/F | Up to 13 weeks
  Apparent clearance of SHR-1819
Pharmacokinetics-Vz/F | Up to 13 weeks
  Apparent volume of distribution during terminal phase of SHR-1819
Pharmacokinetics-t1/2 | Up to 13 weeks
  Terminal elimination half-life of SHR-1819
Change from baseline to end of treatment for TARC/CCL17 | Up to 13 weeks
  TARC/CCL17
Change from baseline to end of treatment for IgE | Up to 13 weeks
  IgE
Immunogenicy of SHR-1819 after administration | Up to 13 weeks
  Anti-drug antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Atridia Pty Limited, Sydney, New South Wales, Australia